CLINICAL TRIAL: NCT06513104
Title: Investigation of the Effect of NNC0519-0130 on the Pharmacokinetics of an Oral Combination Contraceptive (Ethinylestradiol and Levonorgestrel) and Gastric Emptying in Healthy Postmenopausal Females
Brief Title: A Research Study Looking Into the Effect of NNC0519-0130 on Blood Levels of a Birth Control Pill and Emptying of the Stomach in Women After Menopause
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9541-4922; U1111-1294-3433 (Other: World Health Organization (WHO)); 2023-507973-16 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Levonorgestrel; Ethinyl Estradiol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NNC0519-0130 + OC+ paracetamol (Experimental): All participants will initiate treatment with paracetamol (once) and oral contraceptive (Levonorgestrel + Ethinylestradiol) treatment only followed by a period with NNC0519-0130 treatment only, thereafter a period with NNC0519-0130, paracetamol (once) and oral contraceptive treatment.
  Interventions: Drug: NNC0519-0130; Drug: Levonorgestrel + Ethinylestradiol; Drug: Paracetamol

INTERVENTIONS:
Drug: NNC0519-0130 — NNC0519-0130 will be administered subcutaneously.
Drug: Levonorgestrel + Ethinylestradiol — Levonorgestrel + Ethinylestradiol will be administered orally.
Drug: Paracetamol — Paracetamol will be administered orally.

SUMMARY:
The purpose of the study is to investigate if NNC0519-0130 affects the blood levels of a birth control pill that contains the two hormones ethinylestradiol and levonorgestrel. The study will also look into if NNC0519-0130 affects how fast stomach is emptied. Participants will get the new study medicine NNC0519-0130 and will also get birth control pills and paracetamol. The study will last for about 35 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female.
* Age greater than or equal to (≥)45 years at the time of signing informed consent.
* Body weight ≥ 60 kilogram (kg).
* Body mass index (BMI) between 27.0 and 39.9 kilogram per square meter (kg/m^2) (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered to be otherwise healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder, unwillingness or inability which in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol.
* Glycated haemoglobin (HbA1c) ≥ 6.5 percent (%) (48 millimoles per mole (mmol/mol)) at screening.
* Any contraindications for the use of the oral contraception used in the study according to the Microgynon Summary of Product Characteristics, including:

  1. Presence or risk of venous thromboembolism or arterial thromboembolism, e.g., history of migraine with focal neurological symptoms or transitory ischemic attacks.
  2. Undiagnosed vaginal bleeding.
  3. Presence or history of breast cancer.
  4. Presence or history of liver tumours (benign or malignant).
  5. Positive family history of arterial thromboembolism and/or venous thromboembolism (ever in a sibling or parent especially at relatively early age e.g. below 50).
  6. Known hereditary or acquired predisposition for arterial thromboembolism, such as hyperhomocysteinaemia and anti-phospholipid antibodies (anticardiolipinantibodies, lupus anticoagulant).
  7. Known hereditary or acquired predisposition to venous thromboembolism, such as Activated Protein C (APC) resistance (including factor V Leiden), antithrombin III deficiency, protein C deficiency or protein S deficiency.
  8. Dyslipoproteinaemia.
* Use of prescription medicinal products or non-prescription drugs including any herbal medicine known to interfere with the metabolic cytochrome P450 (CYP) pathways, such as hypericum (St. John's Wort), ginseng, garlic, milk thistle, and echinaceae, within 14 days before screening. Exceptions are routine vitamins, occasional use of paracetamol, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation.
* Use of hormone replacement therapy within 4 weeks before screening or intention to initiate treatment with hormone replacement therapy during the study.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Area under the ethinylestradiol plasma concentration time curve during a dosing interval at steady state | Day 8
  Measured in hours picograms per milliliter (h*pg/mL).
Area under the ethinylestradiol plasma concentration time curve during a dosing interval at steady state | Day 188
  Measured in h*pg/mL.
Area under the levonorgestrel plasma concentration time curve during a dosing interval at steady state | Day 8
  Measured in h*pg/mL.
Area under the levonorgestrel plasma concentration time curveduring a dosing interval at steady state | Day 188
  Measured in h*pg/mL.

SECONDARY OUTCOMES:
Maximum ethinylestradiol plasma concentration at steady state | Day 8 and Day 188
  Measured in picograms per milliliter (pg/mL).
Maximum levonorgestrel plasma concentration at steady state | Day 8 and Day 188
  Measured in pg/mL.
Area under the paracetamol concentration-time curve for 0-300 minutes following a standardised meal | Day 1 and Day 181
  Measured in hours micrograms per milliliter (h*μg/mL).
Area under the paracetamol concentration-time curve for 0-60 minutes following a standardised meal | Day 1 and Day 181
  Measured in h*μg/mL.
Maximum paracetamol plasma concentration following a standardised meal | Day 1 and Day 181
  Measured in micrograms per milliliter (μg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com